CLINICAL TRIAL: NCT03940859
Title: Investigation of Dynamic Contrast-Enhanced Magnetic Resonance Imaging Analysis Predicting Prognosis of Intracranial Dissecting Aneurysm With Intramural Hematoma After Endovascular Treatment
Brief Title: Dynamic Contrast-Enhanced Magnetic Resonance Imaging Analysis for Prognosis of Intracranial Dissecting Aneurysm With Intramural Hematoma After Endovascular Treatment
Acronym: DEMAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Principal Investigator, zhangyisen, Attending Doctor of Department of Interventional Neuroradiology, Beijing Neurosurgical Institute
Other Study IDs: NSFC-81801158
Record Dates: First submitted 2019-05-05; First posted 2019-05-07 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Dissecting Aneurysm of Cerebral Artery
Keywords: contrast-enhanced magnetic resonance imaging; intracranial dissecting aneurysm; intramural hematoma; prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DEMAT: Patients with intramural hematoma in intracranial dissecting aneurysm treated by endovascular treatment will be recruited.
  Interventions: Device: intracranial stent, flow diverter and coils

INTERVENTIONS:
Device: intracranial stent, flow diverter and coils — Endovascular treatment was performed under general anesthesia. Patients were treated with internal trapping, stent-assisted coiling or flow diverter as appropriate. After the procedure, patients treated with conventional stent were given 75mg/d clopidogrel for 6 weeks and 100mg/d aspirin for 6months, while patients treated with flow diverter were given 75mg/d clopidogrel for 3 months and 100mg/d aspirin thereafter. All patients were recommended to undergo a 6-month angiographic follow-up.
  Other Names: Low profile Visualized Intraluminal Device (LVIS); Pipeline™(or Flex) Embolization Device(PED)

SUMMARY:
This study will evaluate the feasibility to predict the prognosis of IDA with IMH by DCE-MRI and provide theoretical basis for the prognosis and intervention of the disease.

DETAILED DESCRIPTION:
Intracranial dissecting aneurysm (IDA) was a challenging disease and could result in stroke in young and middle-aged adults. Intramural hematoma, one of the typical imaging findings of IDA, can grow continuously in untreated IDA. Due to relatively high complication rate associated with surgical procedures, endovascular treatments have become the first-line therapy for such lesions. According to whether the parent artery was maintained, endovascular treatment was divided into deconstructive (proximal arterial occlusion and internal trapping) and reconstructive (stent implantation with or without coiling) techniques . However, recanalization of IDA was a great challenge for endovascular treatment and influenced the prognosis of patients.

The formation of an IMH is a critical event in the progress of IDA and IDA may grow because of recurrent IMH even after deconstructive endovascular treatment. Increased IMH size could result in severe compression symptoms or even death. At present, the mechanism of the continuous growth of intramural hematoma after endovascular treatment of IDA is still unclear. Some authors believe that the continuous hemorrhage of the vasa vasorum in the IMH results in the continuous enlargement of the IMH. However, this theory has not been proved by imaging in vivo.

Dynamic contrast-enhanced magnetic resonance imaging analysis for prognosis of intracranial dissecting aneurysm with intramural hematoma after endovascular treatment (DEMAT) is a prospective trial designed to collect a large series of patients with IDAs treated endovascularly to predict the prognosis of IDA with IMH by DCE-MRI and provide theoretical basis for the prognosis and intervention of the disease.

ELIGIBILITY:
Inclusion Criteria:

adult patients (age 18-80 years) patients' ability to cooperate during the MRI examination; patients who are were diagnosed with IDA according to DSA and MRI; expectation of adequate patient safety during these examinations; unequivocal evidence by MRI (IMH>5 mm on the perpendicular plane to the long axis of the vessel) of IDA; IDA treated by the endovascular approach; patients' willingness to participate in the study.

Exclusion Criteria:

patients with pre-existing diagnoses of arteritis, fibromuscular dysplasia, iatrogenic aneurysms or pseudoaneurysms; extracranial dissecting aneurysms extended into the intracranial segment; patients with other diseases or poor general condition with expected survival of less than 2 year; the IDA has already been treated by the endovascular treatment; patients lacking DCE-MRI follow up.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients had an IDA with IMH and received an endovascular treatment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
neovascularization and permeability factors related to enlargement of IMH as assessed by DCE-MRI. | 6 months
  Using DCE-MRI, the parameters as Ktrans and Vp could be calculated and analyzed. These will be studied as a composite indicator for the enlargement of IMH.

SECONDARY OUTCOMES:
clinical factors related to the enlargement of IMH as recorded from medical chart | 6 months
  size, treatment method, device use, follow-up interval, smoke history, hypertension, et al, will be recorded and analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Neurosurgical Institute and Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tian Z, Wang Z, Li W, Zhu W, Liu J, Zhang Y, Yang X, Zhang Y. Dynamic contrast-enhanced MRI analysis for prognosis of intracranial dissecting aneurysm with intramural haematoma after endovascular treatment: an observational registry study. Stroke Vasc Neurol. 2021 Mar;6(1):133-138. doi: 10.1136/svn-2020-000326. Epub 2020 Jul 1. PMID 32611729